CLINICAL TRIAL: NCT00938548
Title: Perioperative Administration of Pregabalin for Pain After Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Severance Hospital, Anesthesia and Pain Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 4-2009-0186
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2009-07

CONDITIONS: Pain, Postoperative
Keywords: mastectomy; pain, postoperative; pregabalin
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients receive oral Placebo 1 hour prior to surgery, and 12 hours later
  Interventions: Drug: Vitamin Complex (placebo)
- Pregabalin (Experimental): Patients receive oral pregabalin 1 hour prior to surgery, and 12 hours later
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 75 mg orally
  Arms: Pregabalin
Drug: Vitamin Complex (placebo) — Vitamin Complex orally
  Arms: Placebo

SUMMARY:
The investigators hypothesize that pregabalin will decrease post-operative pain scores and analgesic use following total mastectomy compared to placebo. The primary outcome will be acute postoperative pain, measured by a verbal numerical rating score (VNRS) and total analgesic consumption during postoperative 48 hours. The secondary outcome will be VNRS at 1 week and 1 month after operation.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesia physical status class I & II
2. Age > 20 and < 70 years
3. Robot- assisted endoscopic thyroidectomy

Exclusion Criteria:

1. Known or suspected allergy, sensitivity, or contraindication to pregabalin or any of the standardized medications
2. Body mass index ≥ 40 kg/m2
3. History of seizure disorder
4. Current therapy with pregabalin, gabapentin, or any opioid
5. Any other physical or psychiatric condition which may impair their ability to cooperate with post-operative study data collection
6. Insulin-dependent diabetes mellitus
7. Renal insufficiency (estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2)

Ages: 21 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia, Seoul, South Korea

REFERENCES:
- [Derived] Kim SY, Song JW, Park B, Park S, An YJ, Shim YH. Pregabalin reduces post-operative pain after mastectomy: a double-blind, randomized, placebo-controlled study. Acta Anaesthesiol Scand. 2011 Mar;55(3):290-6. doi: 10.1111/j.1399-6576.2010.02374.x. PMID 21288209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was approved by the Institutional Ethics Committee of Yonsei University Medical Center.
  Datas were collected between June and December 2009.
Pre-assignment Details: Of a total of 78 patients assessed for eligibility, 70 subjects received pregabalin or placebo after randomization.
  Eight patients were excluded because some patients refused to participate and some patients have psychiatric disorder and insulin-dependent DM.
Period: Overall Study
Arm/Group | Placebo | Pregabalin
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (8) | 51 (9) | 50 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores (Verbal Numerical Rating Scale;VNRS) During Postoperative Hours.
Description: Pain was evaluated using an 11-point verbal numerical rating scale (VNRS). Patients were instructed preoperatively to express their pain on the 0-10 VNRS, where 0 represents no pain at all and 10 represents the worst pain imaginable.
Time Frame: 1, 6, 24, 48 hour
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 35 | 35
Units on a scale
  1 hr | 7 (1.8) [3 to 10] | 5 (2.1) [0 to 9]
  6 hr | 6 (2.1) [2 to 10] | 5 (2.2) [2 to 10]
  24 hr | 5 (1.7) [1 to 8] | 3 (1.5) [1 to 7]
  48 hr | 3 (1.8) [0 to 7] | 2 (1.3) [1 to 5]

2. Primary Outcome: Number of Participants With the Indicated Side Effects - Nausea & Vomiting, Sedation, Headache, Dizziness Etc.
Description: Nausea and vomiting was graded on a four-point scale, where 0 = no nausea, 1 = mild nausea, 2 = severe nausea requiring antiemetics, and 3 = retching and/ or vomiting. Grades 3 and 4 were grouped together as postoperative nausea and vomiting (PONV) and rescue anti-emetic, metoclopramide 10 mg i.v. was given.
Time Frame: 1, 6, 24, 48 hour
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 35 | 35
participants
  PONV | 4 | 3
  sedation | 8 | 13
  headache | 9 | 5
  dizziness | 12 | 17

3. Secondary Outcome: Pain Scores (VNRS) at 1 Week and 1 Month After Operation
Description: as for outcome 1
Time Frame: 1 week, 1 month
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 35 | 35
Units on a scale
  1 week | 2.9 (1.3) | 1.4 (0.9)
  1 month | 1.7 (1.6) | 0.6 (0.6)

ADVERSE EVENTS:
Arm/Group | Placebo | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 18/35 | 19/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | Pregabalin (N=35)
dizziness (Nervous system disorders) | 12 | 17
sedation (Nervous system disorders) | 8 | 13
headache (Nervous system disorders) | 9 | 5
PONV (Gastrointestinal disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No